CLINICAL TRIAL: NCT03920267
Title: A Multi-Center Study to Characterize the Long-Term Safety and Efficacy of BMS-986165 in Subjects With Systemic Lupus Erythematosus
Brief Title: Long-Term Safety and Efficacy Study of Deucravacitinib in Participants With Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM011-074; 2018-003471-35 (EudraCT Number)
Record Dates: First submitted 2019-03-27; First posted 2019-04-18 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — deucravacitinib

STUDY DESIGN:
Intervention Model Description: Participants who successfully complete the protocol-required treatment period of the Phase 2 SLE study (NCT03252587) will be offered the opportunity to continue this study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BMS-986165 Dose 1 (Experimental)
  Interventions: Drug: BMS-986165
- BMS-986165 Dose 2 (Experimental)
  Interventions: Drug: BMS-986165
- BMS-986165 Dose 3 (Experimental)
  Interventions: Drug: BMS-986165

INTERVENTIONS:
Drug: BMS-986165 — Specified dose on specified days
  Other Names: Deucravacitinib

SUMMARY:
The main objective of the trial is to characterize the long-term safety and tolerability of BMS-986165 in subjects with Systemic Lupus Erythematosus (SLE).

ELIGIBILITY:
Inclusion Criteria:

* Completion of SLE Study (NCT03252587) through the protocol-required treatment period, and currently receiving blinded study drug. Note: If a subject is not receiving blinded study drug due to exceptional circumstances (eg, missed investigational product [IP] due to COVID-19 pandemic, delays in study approval, etc), the subject may be allowed to enroll with approval from the BMS Clinical Trial Physician or designee.

Exclusion Criteria:

* Any disease or medical condition that, in the opinion of the investigator, would make the subject unsuitable for this study, would interfere with the interpretation of subject safety or study results, or considered unsuitable by the investigator for any other reason
* Evidence of active tuberculosis (TB)

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Up to 30 days after last treatment dose (approximately 178 weeks)
Number of participants with Serious Adverse Events (SAEs) | Up to 30 days after last treatment dose (approximately 178 weeks)
Number of participants with AEs leading to discontinuation | Up to 30 days after last treatment dose (approximately 178 weeks)
Number of participants with abnormal change from baseline in laboratory measurements over time | Up to 30 days after last treatment dose (approximately 178 weeks)
Number of participants with abnormal change from baseline in vital signs over time | Up to 30 days after last treatment dose (approximately 178 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (98):
- United States (25):
  - Local Institution - 0077, Birmingham, Alabama
  - Local Institution - 0030, El Cajon, California
  - Local Institution - 0049, Torrance, California
  - Local Institution - 0074, New Haven, Connecticut
  - Local Institution - 0115, Aventura, Florida
  - Local Institution - 0044, Brandon, Florida
  - Local Institution - 0140, Gainesville, Florida
  - Local Institution - 0133, Orlando, Florida
  - Local Institution - 0032, Ormond Beach, Florida
  - Local Institution - 0048, Tampa, Florida
  - Local Institution - 0094, Atlanta, Georgia
  - Local Institution - 0050, Lawrenceville, Georgia
  - Local Institution - 0123, Brooklyn, New York
  - Local Institution - 0131, New York, New York
  - Local Institution - 0071, Chapel Hill, North Carolina
  - Local Institution - 0031, Charlotte, North Carolina
  - Local Institution - 0064, Oklahoma City, Oklahoma
  - Local Institution - 0035, Wyomissing, Pennsylvania
  - Local Institution - 0121, Charleston, South Carolina
  - Local Institution - 0001, Jackson, Tennessee
  - Local Institution - 0041, Austin, Texas
  - Tekton Research - Austin, Austin, Texas
  - Local Institution - 0114, Dallas, Texas
  - Local Institution - 0037, Houston, Texas
  - Local Institution - 0046, Mesquite, Texas
- Argentina (7):
  - Clinica Adventista Belgrano, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Local Institution - 0125, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Local Institution - 0098, Rosario, Santa Fe Province
  - Local Institution - 0091, San Miguel de Tucum, Tucumán Province
  - Local Institution - 0100, CABA
  - Local Institution - 0122, Córdoba
  - Local Institution - 0095, Mendoza
- Brazil (7):
  - Local Institution - 0116, Salvador, Estado de Bahia
  - Local Institution - 0118, Goiߡ, Goiás
  - Local Institution - 0106, Juiz de Fora, Minas Gerais
  - Local Institution - 0120, Curitiba, Paraná
  - Local Institution - 0107, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0111, São Bernardo do Campo, São Paulo
  - Local Institution - 0105, São Paulo
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - Local Institution - 0136, Toronto, Ontario
- Colombia (4):
  - Local Institution - 0108, Barranquilla
  - Local Institution - 0101, Bogotá
  - Local Institution - 0103, Chía
  - Local Institution - 0096, Zipaquirá
- Hungary (3):
  - Local Institution - 0039, Debrecen
  - Local Institution - 0038, Gyula
  - Local Institution - 0045, Szeged
- Japan (10):
  - National Hospital Organization Chibahigashi National Hospital, Chiba, Chiba
  - Local Institution - 0092, Kitakyushu, Fukuoka
  - Local Institution - 0119, Sapporo, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Local Institution - 0063, Sendai, Miyagi
  - Local Institution - 0069, Shimotsuke, Tochigi
  - Local Institution - 0065, Chuo-ku, Tokyo
  - Local Institution - 0078, Tokyo
  - Local Institution - 0066, Tokyo
  - Local Institution - 0093, Tokyo
- Mexico (6):
  - Local Institution - 0080, León, Guanajuato
  - Local Institution - 0086, León, Guanajuato
  - Investigacion Biomedica para el Desarrollo de Farmacos S.A. de C.V., Zapopan, Jalisco
  - Local Institution - 0087, Mexico City, Mexico City
  - Local Institution - 0084, Monterrey, Nuevo León
  - Local Institution - 0082, San Luis Potosí City
- Poland (12):
  - Local Institution - 0025, Bydgoszcz
  - Local Institution - 0015, Kościan
  - Local Institution - 0014, Krakow
  - Local Institution - 0027, Krakow
  - Local Institution - 0018, Krakow
  - Local Institution - 0016, Lublin
  - Local Institution - 0024, Poznan
  - Local Institution - 0029, Sosnowiec
  - Local Institution - 0019, Warsaw
  - Local Institution - 0022, Warsaw
  - Local Institution - 0010, Wroclaw
  - Local Institution - 0023, Wroclaw
- Romania (3):
  - Local Institution - 0033, Brasov
  - Local Institution - 0004, Galati
  - Local Institution - 0002, Râmnicu Vâlcea
- Russia (10):
  - Local Institution - 0056, Kemerovo
  - Local Institution - 0072, Novosibirsk
  - Local Institution - 0057, Orenburg
  - Local Institution - 0062, Saint Petersburg
  - Local Institution - 0058, Saint Petersburg
  - Local Institution - 0070, Smolensk
  - Local Institution - 0055, Vladimir
  - Local Institution - 0068, Yaroslavl
  - Local Institution - 0060, Yaroslavl
  - Local Institution - 0061, Yekaterinburg
- South Korea (2):
  - Local Institution, Seoul
  - Local Institution - 0053, Suwon
- Spain (3):
  - Local Institution - 0126, Málaga
  - Local Institution - 0138, Sabadell
  - Local Institution - 0124, Seville
- Taiwan (4):
  - Local Institution - 0052, Taichung
  - Local Institution - 0051, Taipei
  - Local Institution, Taipei
  - Local Institution - 0137, Taipei

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com